CLINICAL TRIAL: NCT01519934
Title: Retrospective Evaluation of the Ulthera System for Lifting and Tightening of the Face and Neck
Brief Title: A Retrospective Study to Evaluate the Effectiveness of the Ulthera System
Status: Completed | Type: Observational
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Other Study IDs: ULT-120
Record Dates: First submitted 2011-11-07; First posted 2012-01-27 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-11

CONDITIONS: Skin Laxity; Wrinkles
Keywords: Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.; Ultrasound treatment for skin tightening
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ulthera-treated subjects: All enrolled subjects will have received an Ulthera treatment prior to enrollment.

SUMMARY:
Up to 120 subjects within the study site's practice who have already had an Ultherapy™ treatment to the face and neck will be enrolled to monitor treatment effectiveness. Follow-up visits will occur at 90 and 180 days post-treatment. Study images will be obtained at each follow-up visit.

DETAILED DESCRIPTION:
This is a retrospective, single-center clinical trial to evaluate the efficacy of the Ulthera System for non-invasive treatment of skin texture and laxity six months after treatment. Global Aesthetic Improvement Scale scores, patient satisfaction questionnaires, and quality of life questionnaires will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 25-85 years.
* Subject in good health.
* Received Ultherapy™ treatment prior to or on October 1, 2011, and must have had pre-treatment baseline photographs taken.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits.
* Absence of physical or psychological conditions unacceptable to the investigator.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Significant scarring in areas treated.
* Open wounds or lesions in the areas treated.
* Severe or cystic acne on the areas treated.
* Inability to understand the protocol or to give informed consent.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of males and females from the investigator's practice between 25 and 85 years of age, who have received an Ultherapy™ treatment on or prior to October 1, 2011, who had pre-treatment baseline photographs taken, and who have chosen to participate in this clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel Goldman, MD, Principal Investigator — Dermatology Cosmetic Laser Associates
Locations (1):
- Dermatology Cosmetic Laser Associates, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who had received an Ulthera treatment to the face and upper neck at two treatment depths at one study site were recruited for study participation.
Groups:
- Ulthera-treated Subjects: All enrolled subjects had received one Ulthera treatment on the face and neck at two treatment depths, 4.5mm and 3.0mm depths, prior to enrollment.
Period: Overall Study
Arm/Group | Ulthera-treated Subjects
Started | 48
Completed | 45
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Subjects who had received a dual depth Ulthera treatment to the face and upper neck prior to enrollment and met all entrance criteria.
Arm/Group | Ulthera-treated Subjects
Number analyzed (Participants) | 48
Age, Continuous [Mean (Full Range); unit: years] | 58 [39 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1
  Caucasian | 42
  Hispanic/Latino | 3
  Native Hawaiian or Other Pacific Islander | 1
  More than one race | 1
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Overall Lifting and Tightening of the Skin
Description: Determined by a masked, qualitative assessment of photographs at 180 days post treatment compared to pre-treatment baseline photographs. A panel of three blinded assessors reviewed pre-treatment and post-treatment photos. Each blinded assessor was provided an identical set of pre-treatment and Day 180 post-treatment photos to assess. The pre/post treatment photos were consistent in lighting, subject positioning and focus. The visit interval of each photo, i.e. pre and post treatment, was NOT marked. Each blinded assessor conducted their assessment independently with no input from another blinded assessor, comparing each set of photos. Each assessor indicated those subjects assessed as improved.
Time Frame: Baseline to 180 days post-treatment
Measure: Number; unit: percentage of participants
Arm/Group | Ulthera-treated Subjects
Number analyzed (Participants) | 45
percentage of participants | 67

2. Secondary Outcome: Overall Aesthetic Improvement
Description: Overall aesthetic improvement was assessed based on a Global Aesthetic Improvement Scale (GAIS) scores; PGAIS completed by a clinician assessor, SGAIS completed by the study subject. The GAIS is 5-point scale (1-5) describing an overall assessment as follows:
  1. = Very Much Improved
  2. = Much Improved
  3. = Improved
  4. = No Change
  5. = Worse
Time Frame: Baseline to 180 days post-treatment
Measure: Number; unit: percentage of participants
Arm/Group | Ulthera-treated Subjects
Number analyzed (Participants) | 45
percentage of participants
  Investigator GAIS | 78
  Subject GAIS | 78

3. Secondary Outcome: Subject Perception of Age
Description: Percentage of subjects rated as "looking younger" as measured using a Subject Perception of Age questionnaire.
Time Frame: Baseline to 180 days post-treatment
Measure: Number; unit: percentage of participants
Arm/Group | Ulthera-treated Subjects
Number analyzed (Participants) | 45
percentage of participants | 60

4. Secondary Outcome: Patient Satisfaction
Description: Percentage of subjects reporting satisfaction as measured using a Patient Satisfaction Questionnaire.
Time Frame: 180 days post-treatment
Measure: Number; unit: percentage of participants
Arm/Group | Ulthera-treated Subjects
Number analyzed (Participants) | 45
percentage of participants | 60

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment to 6 months post-treatment.
Arm/Group | Ulthera-treated Subjects
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No